CLINICAL TRIAL: NCT06380998
Title: Effects of Petroleum Compounds on Psychological Health, Cognitive Functions, and the Possible Ameliorating Effect of Whey Protein in a Sample of Petrol Station Workers in Assiut Governorate
Brief Title: Effects of Petroleum Compounds on Psychological Health and Cognitive Functions
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad Hussien Eisa, Assiut University, Faculty of medicine, Forensic medicine and clinical toxicology department, lecturer assistant, Assiut University
Other Study IDs: EPCPHCFAPAEWPSPSWAG
Record Dates: First submitted 2024-04-16; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Cognitive Deterioration
Keywords: Petroleum compounds; psychological heath; cognitive funtions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — urine samples for BTEX metabolites
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- petrol station workers: Petrol station workers of 2 years duration and in direct contact with petroleum compounds vapours
  Interventions: Dietary Supplement: whey protien

INTERVENTIONS:
Dietary Supplement: whey protien — Whey, the supernatant of yogurt and a byproduct of cheese, is rich in protein and consists of β-lactalbumin, α-lactoglobulin, immunogloblin, bovine serum albumin, and other minor proteins. Whey protein is a globally consumed food material and is well known for its health benefits

SUMMARY:
Over the last decade, awareness of the effects of hydrocarbon fuels on neurodegenerative disorders has increased significantly, as they are ubiquitous environmentally toxic chemicals that affect the central nervous system and result in irreversible neuronal damage, as many hydrocarbons can cross the blood-brain barrier through multiple pathways and cause direct toxicity.

DETAILED DESCRIPTION:
Petrol stations are establishments that retail liquid fuels derived from petroleum, alcohol, and other automotive fuels, with equipment available for their measurement and storage. This process, linked to gasoline distribution, can be a significant source of volatile organic compounds (VOCs), such as benzene, toluene, ethylbenzene, and xylene isomers (BTEX), the primary volatile hydrocarbons derived from petroleum.

Headache, fatigue, dizziness, respiratory tract infections, skin allergies, eye infections, and impairment of memory have been experienced by a few people immediately following exposure to some solvents. CNS depression is a common physiological outcome caused by high exposure to some VOCs. General anaesthetic effects, and as a most severe outcome, unconsciousness and, in some cases, death, may occur at the end.

Long-term exposure to organic solvents may cause permanent central nervous system disturbances, a condition called chronic solvent encephalopathy (CSE).

Cognitive symptoms and neuropsychological signs, or issues with memory, focus, and learning, are the hallmarks of CSE, which is underdiagnosed and characterized by these symptoms as well as possible side effects like headaches, fatigue, balance issues, and mild depression. If exposure stops, though, the illness will not worsen.

We are discovering more about the importance of nutrition and its impact on an individual's susceptibility to illness progression. Diet has been suggested to have an important role in cognitive health and the development of dementia. However, most of the intervention studies conducted to date have mainly assessed the effect of dietary supplements on cognitive function.

The toxicity of inhaled vapours is due to their biotransformation into reactive oxygen species, and several studies have highlighted the capacity of whey protein to increase glutathione (GSH), suggesting that this complex mixture is capable of boosting GSH synthesis, thus reducing oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Workers in direct contact with petroleum compounds in petroleum stations.
* Working for at least 8 continuous hours daily for at least 2 years before enrollment in the study.
* Participants have willingness to participate and have no history for substance abuse

Exclusion Criteria:

* Working for less than 2 years with interrupted exposure.
* The exposure of workers to petroleum compounds is indirect.
* History of psychological and neurodegenerative diseases before starting this job.
* Patients with medical conditions like renal or cardiovascular diseases.
* Individuals with known allergies or contraindications to study supplements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Petrol station workers at Assiut fuel stations with exposure time of 8 continuous hours for at least 2 years
Sampling Method: Non-Probability Sample
Enrollment: 196 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Effects of petroleum compounds on psychological health and cognitive functions of petrol station workers in Assiut | 1 year
  for psychological assessment through symptom check list 90 (revised) and cognitive function through the Mini Mental State Examination (30 points: 25-30: normal; 21-24: mild cognitive impairment; 10-20: moderate; and 0-9: severe) and Wecksler memory scale (higher score indicates better performance, while lower score indicates memory impairment)
To explore the relation between the level of petroleum hydrocarbon metabolites and the severity of psychological heath and cognitive functions disturbance of petrol station workers | 1 year
  urinary metabolites for BTEX through GS-MS
To explore the role of supplements with whey protein in ameliorating these effects | 1 year
  20 g of whey protein 3 times per week for 8 weeks will be given to workers with cognitive difficulties

SECONDARY OUTCOMES:
To assess the relationship between the psychological effects, cognitive functions, and nutritional status of petroleum station workers | 1 year
  relationship between nutritional status, psychological symptoms, and cognitive difficulties through statistics

CONTACTS AND LOCATIONS:
Overall Officials: Safaa M George, professor, Study Director — Assiut University
Locations (1):
- Faculty of medicine, Asyut, Assiut University, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ciulla M, Marinelli L, Cacciatore I, Stefano AD. Role of Dietary Supplements in the Management of Parkinson's Disease. Biomolecules. 2019 Jul 10;9(7):271. doi: 10.3390/biom9070271. PMID 31295842
- [Background] da Silva AT, Machado RP, Martins ML, Dorneles LEG, Dalmarco EM, da Silva EL, Hinnig PF, Wazlawik E. Whey Protein, Vitamins C and E Decrease Interleukin-10 in Chronic Hemodialysis Patients: A Pioneer, Randomized, Double-Blind Pilot Trial. J Ren Nutr. 2024 Jan;34(1):58-67. doi: 10.1053/j.jrn.2023.08.007. Epub 2023 Aug 19. PMID 37598813
- [Background] Furu HM, Sainio M, Hyvarinen HK, Kaukiainen A. Limitations of periodical health examinations in detecting occupational chronic solvent encephalopathy. Occup Environ Med. 2019 Sep;76(9):688-693. doi: 10.1136/oemed-2019-105858. Epub 2019 Jul 18. PMID 31320491
- [Background] Geraldino BR, Nunes RFN, Gomes JB, da Poca KS, Giardini I, Silva PVB, Souza HP, Otero UB, Sarpa M. Evaluation of Exposure to Toluene and Xylene in Gasoline Station Workers. Adv Prev Med. 2021 May 20;2021:5553633. doi: 10.1155/2021/5553633. eCollection 2021. PMID 34104483
- [Background] Gutierrez L, Folch A, Rojas M, Cantero JL, Atienza M, Folch J, Camins A, Ruiz A, Papandreou C, Bullo M. Effects of Nutrition on Cognitive Function in Adults with or without Cognitive Impairment: A Systematic Review of Randomized Controlled Clinical Trials. Nutrients. 2021 Oct 22;13(11):3728. doi: 10.3390/nu13113728. PMID 34835984
- [Background] Sajid Jabbar A, Ali ET. Impact of Petroleum Exposure on Some Hematological Indices, Interleukin-6, and Inflammatory Markers of Workers at Petroleum Stations in Basra City. J Environ Public Health. 2020 Aug 4;2020:7693891. doi: 10.1155/2020/7693891. eCollection 2020. PMID 32831856
- [Background] Kita M, Obara K, Kondo S, Umeda S, Ano Y. Effect of Supplementation of a Whey Peptide Rich in Tryptophan-Tyrosine-Related Peptides on Cognitive Performance in Healthy Adults: A Randomized, Double-Blind, Placebo-Controlled Study. Nutrients. 2018 Jul 13;10(7):899. doi: 10.3390/nu10070899. PMID 30011836